CLINICAL TRIAL: NCT03241602
Title: Multimodal Analgesic Technique for Control of Post-laproscopy Abdominal Pain in Patient Undergoing Diagnostic Gynacological Laproscopy. A Randomized Controlled Trial
Brief Title: Multimodal Analgesic Technique for Control of Post-laproscopy Abdominal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Refaat, lecturer of Anesthiology at faculty of medicine Cairo univeristy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-61-2017
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Decrease Post Laproscopy Shoulder and Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group of Pulmonary recruitment & Intraperitoneal libocai (Active Comparator)
  Interventions: Combination Product: Combined intraperitoneal lidocaine and pulmonary recruitment maneuver
- Group of Intraperitoneal lidocaine (Active Comparator)
  Interventions: Drug: Intraperitoneal lidocaine
- Group of pulmonary recruitment (Active Comparator)
  Interventions: Procedure: Pulmonary Recruitment
- group receive passive exsufflation through port (No Intervention)

INTERVENTIONS:
Drug: Intraperitoneal lidocaine — the investigator prepares syringes 1.75 ml/kg of 0.2% lidocaine (3.5 mg/kg) or the same volume of normal saline, for intraperitoneal administration. The solution to be instillated will be splashed under the right diaphragmatic area by the surgeon and complete the procedure.
  Arms: Group of Intraperitoneal lidocaine
Procedure: Pulmonary Recruitment — pulmonary recruitment maneuver will be done and consist of five manual pulmonary inflations with a maximum pressure of 40 cm H2O. The anestheiologist hold the fifth positive pressure inflation for approximately 5 seconds
  Arms: Group of pulmonary recruitment
Combination Product: Combined intraperitoneal lidocaine and pulmonary recruitment maneuver — the investigator prepares syringes 1.75 ml/kg of 0.2% lidocaine (3.5 mg/kg) or the same volume of normal saline, for intraperitoneal administration. The solution to be instillated will be splashed under the right diaphragmatic area by the surgeon and complete the procedure before the recovery of the patient pulmonary recruitment maneuver will be done and consist of five manual pulmonary inflations with a maximum pressure of 40 cm H2O. The anestheiologist hold the fifth positive pressure inflation for approximately 5 seconds
  Arms: group of Pulmonary recruitment & Intraperitoneal libocai

SUMMARY:
The advancement of laparoscopy and minimal access surgery has greatly influenced the evolution of anaesthetic techniques. However, postoperative pain intensity may be significant, with up to 40% of patients unsatisfied by routine analgesia and up to 80%may require rescue opioids during their hospital stay. Diagnostic gynaecological laparoscopy has no origin of pain other than the abdominal gas insufflations itself only. Pain relief after diagnostic laparoscopy, being a day case, is an issue of great practical importance.The aim of this study is to compare the efficacy of combining both pulmonary recruitment and intraperitoneal lidocaine versus pulmonary recruitment alone to control post - laparoscopy shoulder pain regarding severity and frequency

Study Design :

Interventional Prospective Randomized Double-blind Controlled Trial

Methodology This study is a randomized double blinded control trial. It will be conducted at Kasr-al ainy hospital, faculty of medicine, Cairo university. Approval of ethical committee and written informed consent will be obtained. 88 female patients, aged 18-45 years , ASA 1 or 2 , scheduled for diagnostic gynaecologic laparoscopy will be included. Females who are (ASA) ≥ 3, alcoholic, drug abusers, allergic to amide LAs, with pre-existing chronic pain disorders, or receiving opioids or tranquilizers for > 1 week preoperatively are excluded. Also if the operation included any interventional procedure or was converted to an open procedure, or had postoperative complications that could increase postoperative pain, it will be excluded. Consenting patients will be randomly allocated to either of three study groups : GPL : Patients will receive pulmonary recruitment maneuver and intraperitoneal lidocaine. GPS: Patients will receive pulmonary recruitment maneuver and intraperitoneal saline. GC : Patients will receive passive exsufflation through the port site. The patient will attend at the pre anaesthetic room 1 hour before the procedure. A 20 Gauge cannula will be inserted peripherally and the patient will be premedicated with intravenous Midazolam 0.02 mg kg-1, Ranitidine 50 mg, 10 mg Metoclopramide.

In the operative room, standard monitoring will be applied to the patient. Anaesthesia will be induced with propofol 2 mg kg-1, Fentanyl 1 mcg kg-1 , Atracurium 0.5 mg kg-1 and the trachea will be intubated after mask ventilation for 3 minutes. Anaesthesia will be maintained with IPPV , isoflurane in 100% oxygen and muscular relaxation with atracurium 0.1mg kg-1every 15 minutes. Depth of anaesthesia was adjusted according to clinical signs. Laparoscopy is done using CO2 as distension medium. The patient will be placed in a Trendelenburg position in order to provide optimum conditions for laparoscopic view. In groups GPL and GPS , the investigator prepares syringes 1.75 ml/kg of 0.2% lidocaine (3.5 mg/kg) or the same volume of normal saline, for intraperitoneal administration. This ensures the surgeon and the anaesthesiologist are blind to the patient's group. The solution to be instilled will be splashed under the right diaphragmatic area by the surgeon and complete the procedure. At the end of the procedure, the patient will be placed back from trendelenburg position. In groups GPL and GPS , a pulmonary recruitment maneuver will be done and consist of five manual pulmonary inflations with a maximum pressure of 40 cm H2O. The anesthesiologist hold the fifth positive pressure inflation for approximately 5 seconds. In group GC CO2 will be removed by passive exsufflation through the port site and gentle abdominal pressure will be applied to evacuate the residual gas. Residual neuromuscular block is antagonized with atropine 1.2 mg and neostigmine 2.5 mg and extubation will be done according to extubation criteria. In the recovery room, patient will be asked about post-operative pain and it'll be controlled using Meperidine 1 mg kg-1 and given by a nurse who is unaware of the nature of the intraoperative analgesia. Then, the patient is discharged to the ward according to the standard criteria. In the ward, patient will be asked to fulfill a questionnaire at 6, 8 and 10 hours postoperative using the visual analogue score (VAS) of pain severity. Patients were questioned as to presence of Side effects (nausea, vomiting).

Possible Risk : Pneumothorax , Local anaesthetic toxicity : CNS depression (lightheadedness and dizziness, difficulty focusing, tinnitus, confusion, and circumoral numbness) , excitation ( tremors tonic-clonic convulsions) , respiratory depression and cardiac dysrhythmias .

DETAILED DESCRIPTION:
The advancement of laparoscopy and minimal access surgery has greatly influenced the evolution of anaesthetic techniques. However, postoperative pain intensity may be significant, with up to 40% of patients unsatisfied by routine analgesia and up to 80%may require rescue opioids during their hospital stay. Diagnostic gynaecological laparoscopy has no origin of pain other than the abdominal gas insufflations itself only. Pain relief after diagnostic laparoscopy, being a day case, is an issue of great practical importance. Pain after Laparoscopy is considered to arise from 3 main sources: the incision sites (50% to 70%), the pneumoperitoneum (20% to 30%) in association with both local (peritoneal and diaphragmatic stretching, ischemia, acidosis) and systemic (hypercarbia causing sympathetic nervous system excitation resulting in amplification of the local tissue inflammatory response) changes, and the procedure site (10% to 20%) as postcholecystectomy wound within the liver. Pain can also be referred from the subdiaphragmatic region as shoulder pain. Shoulder pain is often mild in intensity and can remain for 24 hours. Incisional pain is usually mild to moderate in intensity, and maximal immediately postoperatively, subsiding with time. Local anaesthetic (LA) to be filtered preincisional can not entirely eliminate postoperative pain, especially shoulder pain, In contrast, Intraperitoneal local anaesthetic instillation is a known method of providing post-laparoscopy pain relief. Lidocaine is safe and effective in pain relief, improving respiratory functions and early return of bowel motility. The local anaesthetic blocks visceral nociception from the peritoneum locally as well as a having a systemic effect after absorption through the peritoneal surface . The systemic analgesic effect of LA is induced through an anti-inflammatory effect by peripheral suppression of acute chemically induced pain, inhibition of nerve conduction, as well as having a central antihyperalgesic effect. The pulmonary recruitment manoeuvre (RM) can mechanically remove residual carbon dioxide (CO2) after laparoscopic surgery, reduce phrenic nerve irritation, and consequently reduce post-laparoscopic shoulder and upper abdominal pain. The combined effect of these two methods ,using various local anaesthetics , on pain following laparoscopic procedures has not been reported. This study will investigate the efficacy of combining local anaesthetic infiltration of Lidocaine with pulmonary recruitment manoeuvre on postoperative pain following diagnostic Gynaecologic laparoscopy. For blinding, Pulmonary recruitment maneuver will be combined with intraperitoneal instillation of saline. However, intraperitoneal saline is a known simple maneuver to decrease shoulder pain. A possible explanation is that saline displaces residual pockets of gas from within the peritoneal cavity and thereby prevents loss of suction support between the liver and diaphragm. In this study we hypothesized that combining simple maneuver like pulmonary recruitment with intraperitoneal instillation of local anaesthetic would be more effective than pulmonary recruitment alone.

The aim of this study is to compare the efficacy of combining both pulmonary recruitment and intraperitoneal lidocaine versus pulmonary recruitment alone to control post - laparoscopy shoulder pain regarding severity and frequency

Study Design :

Interventional Prospective Randomized Double-blind Controlled Trial

Study Methods

Methodology This study is a randomized double blinded control trial. It will be conducted at Kasr-al ainy hospital, faculty of medicine, Cairo university. Approval of ethical committee and written informed consent will be obtained. 88 female patients, aged 18-45 years , ASA I or II , scheduled for diagnostic gynaecologic laparoscopy will be included. Females who are (ASA) ≥ 3, alcoholic, drug abusers, allergic to amide LAs, with pre-existing chronic pain disorders, or receiving opioids or tranquilizers for > 1 week preoperatively are excluded. Also if the operation included any interventional procedure or was converted to an open procedure, or had postoperative complications that could increase postoperative pain, it will be excluded. Consenting patients will be randomly allocated to either of three study groups : GPL : Patients will receive pulmonary recruitment maneuver and intraperitoneal lidocaine. GPS: Patients will receive pulmonary recruitment maneuver and intraperitoneal saline. GC : Patients will receive passive exsufflation through the port site. The patient will attend at the pre anaesthetic room 1 hour before the procedure. A 20 Gauge cannula will be inserted peripherally and the patient will be premedicated with intravenous Midazolam 0.02 mg kg-1, Ranitidine 50 mg, 10 mg Metoclopramide.

In the operative room, standard monitoring (electrocardiography, pulse oximetry and non-invasive blood pressure measurement) will be applied to the patient.

Anaesthesia will be induced with propofol 2 mg/ kg, Fentanyl 1 mcg/ kg , Atracurium 0.5 mg kg-1 and the trachea will be intubated after mask ventilation for 3 minutes. Anaesthesia will be maintained with IPPV , isoflurane in 100% oxygen and muscular relaxation with atracurium 0.1mg kg-1every 15 minutes. Depth of anaesthesia was adjusted according to clinical signs. Laparoscopy is done using CO2 as distension medium. Veress needle is introduced at first through lower border of umbilicus and water test is done to ensure intraperitoneal placement. Then, reaching proper distension pressure is ensured by disappearance of dullness over lower border of the liver. The pressure will be about 15 mmHg. The patient will be placed in a Trendelenburg position in order to provide optimum conditions for laparoscopic view. A 10 mm laparoscopic trocar is introduced with 45 degree towards pelvis and zero camera is introduced through the cannula trocar. Second puncture can be done through right or left iliac fossae. In groups GPL and GPS , the investigator prepares syringes 1.75 ml/kg of 0.2% lidocaine (3.5 mg/kg) or the same volume of normal saline, for intraperitoneal administration. This ensures the surgeon and the anaesthesiologist are blind to the patient's group. The solution to be instilled will be splashed under the right diaphragmatic area by the surgeon and complete the procedure. At the end of the procedure, the patient will be placed back from trendelenburg position. In groups GPL and GPS , a pulmonary recruitment maneuver will be done and consist of five manual pulmonary inflations with a maximum pressure of 40 cm H2O. The anesthesiologist hold the fifth positive pressure inflation for approximately 5 seconds. In group GC CO2 will be removed by passive exsufflation through the port site and gentle abdominal pressure will be applied to evacuate the residual gas. Residual neuromuscular block is antagonized with atropine 1.2 mg and neostigmine 2.5 mg and extubation will be done according to extubation criteria. In the recovery room, patient will be asked about post-operative pain and it'll be controlled using Meperidine 1 mg/ kg and given by a nurse who is unaware of the nature of the intraoperative analgesia. Then, the patient is discharged to the ward according to the standard criteria. In the ward, patient will be asked to fulfill a questionnaire at 6, 8 and 10 hours postoperative using the visual analogue score (VAS) of pain severity. The patients were asked to complete a 10-cm linear analogue scale for shoulder pain, which ranged from 0 for no pain at all to 10 for the worst pain imaginable. Patients were questioned as to presence of Side effects (nausea, vomiting).

Possible Risk Pneumothorax , Local anaesthetic toxicity : CNS depression (lightheadedness and dizziness, difficulty focusing, tinnitus, confusion, and circumoral numbness) , excitation ( tremors tonic-clonic convulsions) , respiratory depression and cardiac dysrhythmias .

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, aged 18-45 years scheduled for diagnostic Gynaecologic laparoscopy.
2. American Society of Anesthesiology physical status 1 or 2.

Exclusion Criteria:

1. American Society of Anesthesiology (ASA) physical status ≥ 3
2. Allergy or hypersensitivity to amide type local anaesthetics;
3. Pre-existing chronic pain disorders;
4. Receiving opioids or tranquilizers for > 1 week preoperatively;
5. History of alcohol or drug abuse.
6. If the operation included any interventional procedure or was converted to an open procedure, or had postoperative complications that could increase postoperative pain

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — as the selected surgery is diagnostic laparoscopy done only for female as this type of surgery there will be no source of pain other than abdominal distension
Enrollment: 88 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain measuring 6 hours postoperative | 6 hours post-oprative
  post-operative pain measured using Visual Analogue Scale ,The patients were asked to complete a 10-cm linear analogue scale for shoulder pain, which ranged from 0 for no pain at all to 10 for the worst pain imaginable

SECONDARY OUTCOMES:
Post-operative Pain measuring Visual analogue scale 8 and 10 hour | 8 , 10 Hours Post-operative
  questionnaire will done for the patient at 8, 10 hour using VAS
Post-operative Nausea and Vomitting | 2 hours
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine CAIRO UNIVERISTY, Cairo, Egypt